CLINICAL TRIAL: NCT06347614
Title: Modified Radical Prostatectomy for Prostate Cancer Patients With Enlarged Prostate and Severe Lower Urinary Tract Symptoms: a Single-center, Retrospective Study
Acronym: Two-step RP
Status: Active, not recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yonghong Li, Professor, Sun Yat-sen University
Other Study IDs: 2021-FXY-042
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Two-step Radical Prostatectomy
  Interventions: Procedure: Two-step Radical Prostatectomy

INTERVENTIONS:
Procedure: Two-step Radical Prostatectomy — The first step was the enucleation of the hyperplastic adenoma, followed by the anterograde radical prostatectomy of residual tissue

SUMMARY:
The goal of this retrospective, observational study is to preliminarily learn about the safety and efficacy of two-step radical prostatectomy in the treatment of low- to intermediate-risk prostate cancer patients with enlarged prostate and severe benign prostatic hyperplasia. The main questions it aims to answer are: 1. Whether two-step prostatectomy is safe enough to decrease the surgical difficulty of these patients? 2. Whether the oncologic control is promising?

ELIGIBILITY:
Inclusion Criteria:

Diagnosed as prostate cancer pathologically by prostate biopsy Evaluated as localized prostate cancer by imaging studies Prostate volume>70mL evaluated by transrectal ultrasonography or multi-parametric magnetic resonance imaging Gleason score≤ 4+3=7 Preoperative PSA<20ng/mL Estimated survival> 10 years； Informed consent is obtained from the patient

Exclusion Criteria:

The patient has received other therapy including radical radiotherapy, transurethral resection of the prostate, cryoablation, HIFU, etc.

Any contraindication of surgery or anaesthesia

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Male with prostate cancer
Study Population: Low- to intermediate-risk localized prostate patient with enlarged prostate and severe benign prostatic hyperplasia
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Biochemical Recurrence-free Survival | 5 years
  Number of participants who are free of biochemical relapse after a specified duration of time. Biochemical recurrence is measured by PSA levels. Biochemical recurrence was defined as a measurable serum PSA concentration 0.2 ng/ml or greater.

SECONDARY OUTCOMES:
Surgical time | Intraoperative
  Defined as the time duration from the incision at the opening to the end of closing the incision
Estimated blood loss | Intraoperative
  Defined as all the blood loss counting during the surgery
Hospital stay | From date of surgery until the date of discharge, an average of 7 days
  Defined as the time duration between the first day after surgery to the day of discharge
Continence ContinenceContinence Continence Continence Continence Continence Continence Continence Continence | 2 weeks, 1 months, 3 months, 6 months, 12 months after surgery
  Evaluated with the use of pad per day. Using no more than 1 pad per day is defined as complete continence
Lower urinary tract symptoms | 1 months, 3 months, 6 months, 12 months after surgery
  Evaluated with International Prostatic Symptom Score (IPSS). 1-7: Mild 8-19:Moderate 20-35: Severe
Erectile function | 6 months, 12 months and 24 months after surgery
  Evaluated with International Index of Erectile Function-5 (IIEF-5).The IIEF-5 score is the sum of the ordinal responses to the 5 items.
  22-25: No erectile dysfunction 17-21: Mild erectile dysfunction 12-16: Mild to moderate erectile dysfunction 8-11: Moderate erectile dysfunction 5-7: Severe erectile dysfunction
Positive surgical margin rate | Through study completion, an average of 5 year
  Defined as the proportion of patients with positive surgical margin of the whole prostate and the margin between the hyperplastic adenoma and the residual gland evaluated by pathologists. The location of positive margin will be documented.
Complication | Through study completion, an average of 5 year
  All the complications which was evaluated relevant to the surgery will be documented and graded by Clavien-Dindo grade system.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China